CLINICAL TRIAL: NCT01721681
Title: A Phase III Open, Multicentre Study to Investigate the Safety, Pharmacokinetics and Efficacy of BPL's High Purity Factor X in the Prophylaxis of Bleeding in Factor X Deficient Children Under the Age of 12 Years
Brief Title: A Study to Investigate Bio Product Laboratory Ltd (BPL's) Factor X in the Prophylaxis of Bleeding in Children <12 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Ten 02; 2012-003093-98 (EudraCT Number)
Record Dates: First submitted 2012-10-25; First posted 2012-11-06 (Estimated); Results first posted 2018-03-07 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Factor X Deficiency
MeSH Terms: conditions — Factor X Deficiency | interventions — Factor X

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FACTOR X (Experimental): At the Baseline Visit, eligible children will receive a bolus dose of 50 IU/kg FACTOR X. After the Baseline Visit, children will be treated with FACTOR X prophylactically for a period of 6 months (26 weeks).
  A dosing regimen of 40-50 IU/kg twice a week is recommended, but is not mandatory. Each dose of FACTOR X must not exceed 60 IU/kg.
  Interventions: Biological: FACTOR X

INTERVENTIONS:
Biological: FACTOR X

SUMMARY:
The primary objective of the study is to assess the efficacy of FACTOR X in the prevention of bleeding when given as routine prophylaxis over 12 months.

The secondary objectives of the study are:

1. To assess the pharmacokinetics of FACTOR X after a single dose of 50 IU/kg.
2. To assess the safety of FACTOR X when given as routine prophylaxis over 6 months (26 weeks).

ELIGIBILITY:
Inclusion Criteria

1. Children with hereditary severe or moderate FX deficiency (FX:C <5 IU/dL), based on their lowest reliable FX:C recorded.
2. Children under 12 years old, whose parent/guardian has given informed consent.
3. Children with a history of severe bleeding e.g.: intracranial haemorrhage, before starting prophylactic therapy, OR a mutation in the F10 gene causing a documented severe bleeding phenotype.

Exclusion Criteria

1. Children must not suffer from clinically significant liver disease, renal disease, or other coagulopathy or thrombophilia
2. Children must have no history or suspicion of inhibitors to factor X.
3. Children who have known or suspected hypersensitivity to the investigational medicinal product or its excipients.
4. Children with a history of unreliability or non-cooperation.
5. Children who are participating or have taken part in another trial within the last 30 days.
6. Children planning more than 4 weeks' continuous absence from the locality of the investigational site, between the Screening Visit and the End of Study Visit at approximately 6 months (26 weeks) post-Baseline.

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2015-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ri Liesner, Dr, Principal Investigator — Great Ormond Street Hospital
Locations (3):
- United Kingdom (3):
  - Addenbrookes Hospital, Cambridge
  - Great Ormond Street Hospital, London
  - Sheffield Children's Hospital, Sheffield

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two subjects completed less than 26 weeks in the study. The subjects were re-enrolled and data from their first treatment cycle was excluded from the per-protocol analysis. 9 unique subjects were enrolled event though there were 11 treatment cycles.
Groups:
- Overall Study: At the Baseline Visit, eligible children received a bolus dose of 50 IU/kg FACTOR X. After the Baseline Visit, children were treated with FACTOR X prophylactically for a period of 6 months (26 weeks).
  A dosing regimen of 40-50 IU/kg twice a week was recommended, but was not mandatory. Each dose of FACTOR X was not to not exceed 60 IU/kg.
Period: Overall Study
Arm/Group | Overall Study
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Human Coagulation FACTOR X: At the Baseline Visit, eligible children received a bolus dose of 50 IU/kg FACTOR X. After the Baseline Visit, children were treated with FACTOR X prophylactically for a period of 6 months (26 weeks).
  A dosing regimen of 40-50 IU/kg twice a week was recommended, but was not mandatory. Each dose of FACTOR X was not to not exceed 60 IU/kg.
Arm/Group | Human Coagulation FACTOR X
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Region of Enrollment [Number; unit: participants]
  United Kingdom | 9

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Excellent Reduction in Bleeding When Given FACTOR X as Routine Prophylaxis Over 6 Months
Description: The Investigator's assessment of the efficacy of FACTOR X in reduction/prevention of bleeding when given as routine prophylaxis over 6 months.
  The efficacy was assessed according to tabulated criteria; Excellent, good, poor, unassessable.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants | 9

2. Secondary Outcome: Safety of FACTOR X: Number of Participants Experiencing Adverse Events
Description: One of the secondary objectives was to assess the safety of FACTOR X when given as routine prophylaxis over 6 months (26 weeks). The general strategy of the safety evaluation was to examine the summaries for any trends. No formal hypothesis was carried out. The number of participants who experienced Adverse Events is provided.
Time Frame: 6 months
Population: The safety evaluation examined the summaries for any trends. No formal hypothesis was carried out.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants | 8

3. Secondary Outcome: Pharmacokinetics: FX:C Incremental Recovery
Description: One of the secondary objectives was to assess the pharmacokinetics (FX:C incremental recovery 30 minute post-dose at the Visit 1 (Baseline) and the End of Study Visit after a single dose of 50 IU/kg). The overall mean IR calculated for both visits is presented in the outcome measure table.
Time Frame: Baseline Visit and End of Study Visit, 30 minutes post-dose
Population: Plasma concentrations were obtained for FX:C for all 9 subjects at 30 minutes post dose at Visit 1 and Visit 5.
Measure: Mean (95% Confidence Interval); unit: IU/dL
Arm/Group | Overall Study
Number analyzed (Participants) | 9
IU/dL | 1.74 [1.66 to 1.82]

ADVERSE EVENTS:
Time Frame: From signing of informed consent form until 28 days post-last dose. For subjects who had received FACTOR X on compassionate use prior to study entry, retrospective adverse events data was collected as part of medical history.
Arm/Group | Human Coagulation FACTOR X
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 3/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human Coagulation FACTOR X (N=9)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1)
Influenza A (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human Coagulation FACTOR X (N=9)
Parvovirus IgM, no symptoms (Investigations) | 1 (1)
Pain In Back Of Leg (Musculoskeletal and connective tissue disorders) | 1 (2)
Aneamia (Blood and lymphatic system disorders) | 3 (3)
Intermittent Low Grade Fever (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
High Temperature/Fever (General disorders) | 3 (5)
Headache (Nervous system disorders) | 2 (2)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1)
Cold (Infections and infestations) | 3 (4)
Increased Temperature (Investigations) | 1 (1)
Viral Infection (Infections and infestations) | 2 (2)
Chest Infection (Infections and infestations) | 1 (2)
Wheeze (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (2)
Positive MRSA Swab To Groin (Infections and infestations) | 1 (1)
Pain In Left Arm (Musculoskeletal and connective tissue disorders) | 1 (1)
Influenza A (Infections and infestations) | 1 (1)
Coryzal (Infections and infestations) | 2 (2)
Lethargy (Nervous system disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
2 subjects completed less than 26 weeks in the study. The subjects were re-enrolled and data from their first treatment cycle was excluded from the Per-Protocol analysis. 9 unique subjects were enrolled even though there were 11 treatment cycles

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days